CLINICAL TRIAL: NCT07115459
Title: Protocol for Developing and Validating a Multimodal Brain Monitoring-Based Prognostic Model for Neurocritical Patients: A Prospective, Observational, Multicenter Cohort Study
Brief Title: Development and Validation of a Prognostic Model for Neurocritical Patients Using Multimodal Brain Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Changsha Fourth Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024070747-2
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Acute Brain Injury Coma; Neurocritical Care; Cerebral Infarction; Intracranial Hemorrhages; Subarachnoid Hemorrhage; Severe Traumatic Brain Injury
Keywords: Multimodal Brain Monitoring; Prognostic Model
MeSH Terms: conditions — Cerebral Infarction; Intracranial Hemorrhages; Subarachnoid Hemorrhage; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate a prognostic model for neurocritical patients using multimodal brain monitoring data. By combining data from various monitoring techniques such as EEG, TCD, and NIRS, this model will help predict 90-day outcomes (awake, comatose, or deceased) and support personalized treatment decisions. The study is observational and involves no experimental interventions.

DETAILED DESCRIPTION:
This study is a prospective, observational, multicenter cohort study conducted in China. It focuses on neurocritical patients with acute brain injury, including large cerebral infarction, intracranial hemorrhage, subarachnoid hemorrhage, or severe traumatic brain injury. The study will collect multimodal data from EEG, TCD, and NIRS monitoring within 1-3 days of ICU admission. Machine learning algorithms will be used to develop a model predicting 90-day outcomes, categorized as awake, comatose, or deceased. The study population includes patients aged 18-80 years. Exclusion criteria include pre-existing severe neurological disorders, incomplete monitoring data, or withdrawal during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years, no gender restrictions.
2. Diagnosed with acute brain injury (ABI), including one of the following: large cerebral infarction, supratentorial large-volume intracerebral hemorrhage, subarachnoid hemorrhage, or severe traumatic brain injury, with imaging evidence (CT or MRI) supporting the diagnosis.
3. On ICU admission, Glasgow Coma Scale (GCS) eye response = 1 (no eye opening) and motor score ≤ 5 (does not follow commands); or within 48 hours, neurological deterioration with no eye opening and motor score reduced to ≤ 5 (total GCS score ≤ 8).
4. Able to undergo continuous multimodal monitoring, with an expected ICU stay of ≥72 hours.
5. Informed consent signed by the family or legal representative.

Exclusion Criteria:

1. Confirmed brain death on admission or imaging showing irreversible brain herniation.
2. Severe trauma unrelated to brain injury (e.g., multiple fractures, spinal cord injuries, or visceral rupture) that may interfere with brain function monitoring or outcome assessment.
3. Pre-existing severe neurological disorders such as epilepsy, severe encephalopathy, or chronic intracranial conditions (e.g., brain tumors or hydrocephalus).
4. Inability to perform multimodal monitoring due to technical issues (e.g., equipment failure or sensor installation problems).
5. Predicted survival time <24 hours after admission, or family members choose to withdraw treatment.
6. Refusal to participate in the study by the patient or their legal representative.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurocritical patients aged 18-80 years with acute brain injury admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
90-day Outcome Prediction | 90-day
  The primary outcome is the prediction of patient status at 90 days post-ICU admission, categorized as awake, comatose, or deceased.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to privacy, ethical, or regulatory considerations